CLINICAL TRIAL: NCT01488669
Title: Robot Assisted Supraomohyoid Neck Dissection Via Retroauricular Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2011-0005
Record Dates: First submitted 2011-12-05; First posted 2011-12-08 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Head and Neck Neoplasms
Keywords: head and neck neoplasms; neck dissection; robotics
MeSH Terms: conditions — Head and Neck Neoplasms

ARMS (2):
- Robotic neck dissection (Experimental): Robotic neck dissection was performed via modified face lift or retroauricular approach using the robotic arms, while conventional neck dissection was conducted after transverse skin incision from the mastoid tip to the midline.
  Interventions: Procedure: robot assisted neck dissection via retroauricular approach
- Conventional neck dissection (Active Comparator): Neck dissection is performed after an external transverse skin incision.
  Interventions: Procedure: Conventional neck dissection

INTERVENTIONS:
Procedure: robot assisted neck dissection via retroauricular approach — A modified face lift or retroauricular incision is made and subplatysmal skin flap is elevated.The marginal mandibular branch of the facial nerve and spinal accessory nerve is identified and lateral part of level II and III is dissected under direct vision using conventional technique. Then, the robotic arms are inserted and the remaining fibrofatty tissue of level I,II,III are dissected under 3D vision.
  Arms: Robotic neck dissection
Procedure: Conventional neck dissection — A transverse skin incision from the mastoid tip to the midline 2 finger below the mandible is made and subplatysmal skin flap is elevated. The fibrofatty tissue of level I,II,III is dissected while preserving the marginal branch of the facial nerve and the spinal accessory nerve. The vessels are ligated using the conventional tie technique and the Harmonic scalpel.
  Arms: Conventional neck dissection

SUMMARY:
In this study we introduce and evaluate the feasibility of our surgical technique to hide the external scar of neck dissection using the robotic system via a modified facelift or retroauricular approach.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as squamous cell carcinoma of the oral cavity
* no clinically identified cervical lymph node metastasis
* surgery as initial treatment

Exclusion Criteria:

* suspicious neck metastasis
* radiation or chemotherapy before the surgery
* past history of neck surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Number of Retrieved lymph nodes | when the pathologist examine the specimen which is within 1 week after operation
  Number of Retrieved lymph nodes counted from the dissected lymphofatty tissues of the specimen

SECONDARY OUTCOMES:
amount and duration of drainage | daily, 6AM, until the drain is removed at an expected average of 5 days
  the amount of drain (ml)is checked from the closed drain bottle.
length of hospital stay | when the patient leaves the hospital at an an expected average of 9 days
  length of hospital stay (day)
satisfaction score | 3 months after operation
  satisfaction score (from 1 to 5) is evaluated at the out-patient department
  (1 = extremely dissatisfied, 2 = dissatisfied, 3 = average, 4 = satisfied, 5 = extremely satisfied)
Operation time | when the dissected specimen is removed from the patient at the average of 78 min for conventional group and 157 min for robot-assisted group
  Operation time (minutes) from skin incision to the time point of removing the dissected specimen from the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Severance Hospital, Seoul, South Korea

REFERENCES:
- [Background] Song CM, Jung YH, Sung MW, Kim KH. Endoscopic resection of the submandibular gland via a hairline incision: a new surgical approach. Laryngoscope. 2010 May;120(5):970-4. doi: 10.1002/lary.20865. PMID 20422693
- [Background] Roh JL. Retroauricular hairline incision for removal of upper neck masses. Laryngoscope. 2005 Dec;115(12):2161-6. doi: 10.1097/01.MLG.0000181496.22493.5A. PMID 16369160
- [Background] Rodrigo JP, Shah JP, Silver CE, Medina JE, Takes RP, Robbins KT, Rinaldo A, Werner JA, Ferlito A. Management of the clinically negative neck in early-stage head and neck cancers after transoral resection. Head Neck. 2011 Aug;33(8):1210-9. doi: 10.1002/hed.21505. Epub 2010 Dec 6. PMID 21755564
- [Background] Wei WI, Ferlito A, Rinaldo A, Gourin CG, Lowry J, Ho WK, Leemans CR, Shaha AR, Suarez C, Clayman GL, Robbins KT, Bradley PJ, Silver CE. Management of the N0 neck--reference or preference. Oral Oncol. 2006 Feb;42(2):115-22. doi: 10.1016/j.oraloncology.2005.04.006. Epub 2005 Jun 24. PMID 15979931
- [Background] Pitman KT. Rationale for elective neck dissection. Am J Otolaryngol. 2000 Jan-Feb;21(1):31-7. doi: 10.1016/s0196-0709(00)80121-0. No abstract available. PMID 10668674
- [Background] Bailey BJ. Selective neck dissection: the challenge of occult metastases. Arch Otolaryngol Head Neck Surg. 1998 Mar;124(3):353. No abstract available. PMID 9525526
- [Background] Ferlito A, Rinaldo A, Silver CE, Robbins KT, Medina JE, Rodrigo JP, Shaha AR, Takes RP, Bradley PJ. Neck dissection for laryngeal cancer. J Am Coll Surg. 2008 Oct;207(4):587-93. doi: 10.1016/j.jamcollsurg.2008.06.337. Epub 2008 Aug 5. No abstract available. PMID 18926464
- [Background] Pentenero M, Gandolfo S, Carrozzo M. Importance of tumor thickness and depth of invasion in nodal involvement and prognosis of oral squamous cell carcinoma: a review of the literature. Head Neck. 2005 Dec;27(12):1080-91. doi: 10.1002/hed.20275. PMID 16240329
- [Background] Terris DJ, Tuffo KM, Fee WE Jr. Modified facelift incision for parotidectomy. J Laryngol Otol. 1994 Jul;108(7):574-8. doi: 10.1017/s002221510012746x. PMID 7930893
- [Background] Terris DJ, Singer MC, Seybt MW. Robotic facelift thyroidectomy: II. Clinical feasibility and safety. Laryngoscope. 2011 Aug;121(8):1636-41. doi: 10.1002/lary.21832. Epub 2011 Jun 30. PMID 21721012
- [Background] Civantos FJ, Stoeckli SJ, Takes RP, Woolgar JA, de Bree R, Paleri V, Devaney KO, Rinaldo A, Silver CE, Mondin V, Werner JA, Ferlito A. What is the role of sentinel lymph node biopsy in the management of oral cancer in 2010? Eur Arch Otorhinolaryngol. 2010 Jun;267(6):839-44. doi: 10.1007/s00405-010-1215-1. Epub 2010 Mar 5. No abstract available. PMID 20204392
- [Result] Fasunla AJ, Greene BH, Timmesfeld N, Wiegand S, Werner JA, Sesterhenn AM. A meta-analysis of the randomized controlled trials on elective neck dissection versus therapeutic neck dissection in oral cavity cancers with clinically node-negative neck. Oral Oncol. 2011 May;47(5):320-4. doi: 10.1016/j.oraloncology.2011.03.009. Epub 2011 Apr 2. PMID 21459661
- [Result] Shiboski CH, Schmidt BL, Jordan RC. Tongue and tonsil carcinoma: increasing trends in the U.S. population ages 20-44 years. Cancer. 2005 May 1;103(9):1843-9. doi: 10.1002/cncr.20998. PMID 15772957
- [Result] Kang SW, Lee SH, Ryu HR, Lee KY, Jeong JJ, Nam KH, Chung WY, Park CS. Initial experience with robot-assisted modified radical neck dissection for the management of thyroid carcinoma with lateral neck node metastasis. Surgery. 2010 Dec;148(6):1214-21. doi: 10.1016/j.surg.2010.09.016. PMID 21134554